CLINICAL TRIAL: NCT05181254
Title: HEAlth Dialogues for Patients With Mental Illness in Primary Care
Acronym: HEAD-MIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-10-28
Record Dates: First submitted 2021-10-31; First posted 2022-01-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mental Illness; Stress; Fatigue; Sleep Disorder; Depression; Diabetes; Myocardial Disease; Stroke; Death
Keywords: primary health care; health dialogue; long-term follow-up; mental illness
MeSH Terms: conditions — Mental Disorders; Fatigue; Sleep Wake Disorders; Depression; Diabetes Mellitus; Cardiomyopathies; Stroke; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health dialogue (Experimental): Patients > 18 years old seeking primary care for mental illness (depression, anxiety, sleep disorders or stress related problems) will be followed at 12 and 24 months from baseline in a first assessment, and after 5 and 10 years with follow-up in national registers in a later phase. The patient will fill out a web-based questionnaire about lifestyle habits before the visit to the health center and will be called for blood sampling and measurement of blood pressure and BMI. A nurse with special training in the Health Dialogue then meets the patient and provides individually tailored advice based on the patient's unique conditions and the risk profile on the Health Dialogue, such as help with smoking cessation, physical activity on prescription (PaR-S), contact with a dietitian, physiotherapist. A continued contact with a psychologist or physician will be planned if necessary
  Interventions: Behavioral: health dialogue

INTERVENTIONS:
Behavioral: health dialogue — The visual health assessment formulary is based on detailed questions about food, physical activity, heredity, smoking, alcohol, stress and mental illness and measurements such as BMI, blood pressure and blood fats. Patients fill in a web-based questionnaire resulting in a visual colorful scale showing a risk assessment (Figure 1). The Health Dialogue is a prognostic tool that provides an estimate of the increase in risk with current lifestyle habits. The use has shown improvement of lifestyle habits such as smoking cessation, lower intake of fat and higher physical activity level as well as reduced mortality in a long-term follow-up.
  Other Names: The health curve

SUMMARY:
In the current project, primary health care patients with mental illness such as anxiety, depression, fatigue or sleep disorders will be followed. The study includes both health conversations with the health curve as a systematic work with lifestyle habits, and the biochemical risk marker copeptin with a focus on improved lifestyle habits and the development of cardiovascular complications. Participants will be followed up at 12 and 24 months with renewed health interview including the health curve and blood sampling. National registries will be used for a, up to 20 year long follow-up regarding cardiovascular complications and mortality.

DETAILED DESCRIPTION:
Patients with mental illness have an increased risk of cardiovascular morbidity and mortality compared to the rest of the population, partly related to unhealthy lifestyle habits. However, not all risk factors for developing cardiovascular disease are known yet. The interest in studies about the importance of copeptin as a biochemical risk factors has increased in recent years.

Objectives:

The main aim with this project is assessment of the effect of Health Dialogue with the health curve (in swedish; Hälsokurvan) on lifestyle habits and cardiovascular risk factors in patients with mental illness in primary care. The second aim is to assess copeptin's prognostic value and to collect blood samples in a biobank for future research on molecular biomarkers with prognostic value for cardiovascular disease.

Work plan:

The study has a prospective observational design. The method with Health Dialogues is previously validated in a Swedish context and is based on a detailed lifestyle questionnaire, blood testing and personalized counselling by a trained health care professional. The patients will be followed with a new Health Dialogue and blood samples after 12 and 24 months and for 20 years with National Registers

Significance:

The effect of Health Dialogues in patients with mental illness is not studied yet. The current fast implementation of the method in the primary care in south of Sweden (the region of Scania) provides a unique opportunity to study this patient group and the expected benefits of Health Dialogues in the long term, to study a potentially useful risk biomarker (copeptin) as well as to build a biobank for future studies on cardiovascular prognostic risk markers.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old seeking primary care for mental illness (depression, anxiety, sleep disorders or stress related problems

Exclusion Criteria:

* Dementia, not speaking, writing or understanding spoken the Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who change their risk profile | 24 months from baseline
  Proportion of patients who achieve a change in the risk profile on the Health Dialogue. A positive change ("yes") is defined if a larger number of the variables on the Health Curve have improved than deteriorated. "No" is defined as no change or negative change has taken place.

SECONDARY OUTCOMES:
Self reported risk change | At 12 and 24 months from baseline
  Proportion of patients who had change between baseline and follow-up in self-reported lifestyle risk assessment
Proportion of smokers and number of cigarettes per day | At baseline and follow-up at 12 and 24 months from baseline.
  Proportion of patients, self-reported answers about smoking, Yes (number of cigarettes per day) no, or former
Referral to smoking cessation | At 12 and 24 months from baseline
  Proportion of patients who have undergone smoking cessation
Time and intensity in physical activity | At baseline and follow-up at 12 and 24 months from baseline.
  Proportion of patients in number of minutes self-reported in physical activity per week in different intensity
Referral PaR-S | At 12 and 24 months from baseline
  Proportion of patients who have received PaR-S
Referral physiotherapist | At 12 and 24 months from baseline
  Proportion of patients who have received referral to physiotherapist
Alcohol consumption | At baseline and follow-up at 12 and 24 months from baseline.
  Proportion of patients, self-reported number of glasses with 4 cl 40% alcohol per week
Metabolic markers | At 12 and 24 months from baseline
  Overnight fasting venous blood sampling. Change in mmol/L from baseline to follow-up of metabolic markers; total cholesterol, triglycerides, high density lipids (HDL), and low density lipids (LDL)
Referral dietitian | At 12 and 24 months from baseline
  Proportion of patients who have received referral to dietitian
Proportion lost to follow-up | At 12 and 24 months from baseline
  Proportion of dropouts / missed follow-ups
Proportion of patients affected with type 2 diabetes | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected of type 2 diabetes: Diagnosis and date of onset of type 2 diabetes mellitus (ICD 10: E11).
Proportion of patients affected with myocardial infarction | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected with myocardial infarction: Diagnosis and date of onset of myocardial infarction (MI) (I21)
Proportion of patients affected with ischemic stroke | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected of ischemic stroke: Diagnosis and date of onset of ischemic stroke (I63)
Proportion of deaths | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients. Diagnosis and date of death
Proportion of cardiovascular death | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected of cardiovascular death: Diagnosis and date of onset of death, cardiovascular death (ICD 10: I)
Proportion of patients affected with venous thromboembolism | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected of : Diagnosis and date of onset of venous thromboembolism (I82.0-I82.3, I82.8, I82.9 & I82.8W)
Proportion of patients affected by MACE (Myocardial infarction, stroke or cardiovascular death) | From baseline and up to 20 years follow-up
  Long time follow-up in registers. Proportion of patients affected of Myocardial infarction, stroke or cardiovascular death (MACE) up to 20 years from baseline: Diagnosis and date of first onset of ischemic stroke (I63), death, cardiovascular death (ICD 10: I), combined to the composite outcome measure MACE (MI, stroke or cardiovascular death).
Co-peptin | At baseline and follow-up at 12 and 24 months from baseline.
  Measured at baseline in pmol/L. Blood sampling after overnight fasting.
Blood glucose | At baseline and follow-up at 12 and 24 months from baseline.
  Fasting blood glucose from venous blood sampling in mmol/L
BMI | At baseline and follow-up at 12 and 24 months from baseline.
  BMI (weight and height will be combined to report BMI in kg/m^2)
Waist hip ratio (WHR) | At baseline and follow-up at 12 and 24 months from baseline.
  WHR will be calculated by the ratio between waist in cm and and hip in cm
Blood pressure | At baseline and follow-up at 12 and 24 months from baseline.
  Measured (mmHg), sitting at right arm after 10 minutes of resting with both feet on the floor.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Pikkemaat, PhD, Study Chair — Lund University/ Region Skane
Locations (1):
- Peter Nymberg, Helsingborg, Region Skane, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson M, Carek PJ, Sullivan B. Treatment of co-morbid mental illness in primary care: how to minimize weight gain, diabetes, and metabolic syndrome. Int J Psychiatry Med. 2011;41(2):127-42. doi: 10.2190/PM.41.2.c. PMID 21675345
- [Background] Jao NC, Robinson LD, Kelly PJ, Ciecierski CC, Hitsman B. Unhealthy behavior clustering and mental health status in United States college students. J Am Coll Health. 2019 Nov-Dec;67(8):790-800. doi: 10.1080/07448481.2018.1515744. Epub 2018 Nov 28. PMID 30485154
- [Background] Wu Q, Kling JM. Depression and the Risk of Myocardial Infarction and Coronary Death: A Meta-Analysis of Prospective Cohort Studies. Medicine (Baltimore). 2016 Feb;95(6):e2815. doi: 10.1097/MD.0000000000002815. PMID 26871852
- [Background] Bonow RO. Primary prevention of cardiovascular disease: a call to action. Circulation. 2002 Dec 17;106(25):3140-1. doi: 10.1161/01.cir.0000048067.86569.e1. No abstract available. PMID 12485965
- [Background] Stumbo SP, Yarborough BJH, Yarborough MT, Green CA. Perspectives on Providing And Receiving Preventive Health Care From Primary Care Providers and Their Patients With Mental Illnesses. Am J Health Promot. 2018 Nov;32(8):1730-1739. doi: 10.1177/0890117118763233. Epub 2018 Apr 15. PMID 29658287
- [Background] Neeleman J, Oldehinkel AJ, Ormel J. Positive life change and remission of non-psychotic mental illness. A competing outcomes approach. J Affect Disord. 2003 Sep;76(1-3):69-78. doi: 10.1016/s0165-0327(02)00068-x. PMID 12943935
- [Background] Ronngren Y, Bjork A, Kristiansen L, Haage D, Enmarker I, Audulv A. Meeting the needs? Perceived support of a nurse-led lifestyle programme for young adults with mental illness in a primary health-care setting. Int J Ment Health Nurs. 2018 Feb;27(1):390-399. doi: 10.1111/inm.12333. Epub 2017 Apr 4. PMID 28374967
- [Background] Forsyth A, Deane FP, Williams P. A lifestyle intervention for primary care patients with depression and anxiety: A randomised controlled trial. Psychiatry Res. 2015 Dec 15;230(2):537-44. doi: 10.1016/j.psychres.2015.10.001. Epub 2015 Oct 3. PMID 26453120
- [Background] Lingfors H, Persson LG, Lindstrom K, Bengtsson C, Lissner L. Effects of a global health and risk assessment tool for prevention of ischemic heart disease in an individual health dialogue compared with a community health strategy only results from the Live for Life health promotion programme. Prev Med. 2009 Jan;48(1):20-4. doi: 10.1016/j.ypmed.2008.10.009. Epub 2008 Nov 1. PMID 19013188
- [Background] Farnkvist L, Olofsson N, Weinehall L. Did a health dialogue matter? Self-reported cardiovascular disease and diabetes 11 years after health screening. Scand J Prim Health Care. 2008;26(3):135-9. doi: 10.1080/02813430802113029. PMID 18609252
- [Background] Persson LG, Lindstrom K, Lingfors H, Bengtsson C, Lissner L. Cardiovascular risk during early adult life. Risk markers among participants in "Live for Life" health promotion programme in Sweden. J Epidemiol Community Health. 1998 Jul;52(7):425-32. doi: 10.1136/jech.52.7.425. PMID 9799876
- [Background] Lingfors H, Lindstrom K, Persson LG, Bengtsson C, Lissner L. Lifestyle changes after a health dialogue. Results from the Live for Life health promotion programme. Scand J Prim Health Care. 2003 Dec;21(4):248-52. doi: 10.1080/02813430310003282. PMID 14695077
- [Background] Persson LG, Lingfors H, Nilsson M, Molstad S. The possibility of lifestyle and biological risk markers to predict morbidity and mortality in a cohort of young men after 26 years follow-up. BMJ Open. 2015 May 6;5(5):e006798. doi: 10.1136/bmjopen-2014-006798. PMID 25948404
- [Background] Lingfors H, Persson LG. All-cause mortality among young men 24-26 years after a lifestyle health dialogue in a Swedish primary care setting: a longitudinal follow-up register study. BMJ Open. 2019 Jan 29;9(1):e022474. doi: 10.1136/bmjopen-2018-022474. PMID 30696668
- [Background] Enhorning S, Wang TJ, Nilsson PM, Almgren P, Hedblad B, Berglund G, Struck J, Morgenthaler NG, Bergmann A, Lindholm E, Groop L, Lyssenko V, Orho-Melander M, Newton-Cheh C, Melander O. Plasma copeptin and the risk of diabetes mellitus. Circulation. 2010 May 18;121(19):2102-8. doi: 10.1161/CIRCULATIONAHA.109.909663. Epub 2010 May 3. PMID 20439785
- [Background] Tasevska I, Enhorning S, Persson M, Nilsson PM, Melander O. Copeptin predicts coronary artery disease cardiovascular and total mortality. Heart. 2016 Jan;102(2):127-32. doi: 10.1136/heartjnl-2015-308183. Epub 2015 Dec 9. PMID 26661323
- [Background] Enhorning S, Christensson A, Melander O. Plasma copeptin as a predictor of kidney disease. Nephrol Dial Transplant. 2019 Jan 1;34(1):74-82. doi: 10.1093/ndt/gfy017. PMID 29471407
- [Background] Pikkemaat M, Melander O, Bengtsson Bostrom K. Association between copeptin and declining glomerular filtration rate in people with newly diagnosed diabetes. The Skaraborg Diabetes Register. J Diabetes Complications. 2015 Nov-Dec;29(8):1062-5. doi: 10.1016/j.jdiacomp.2015.07.006. Epub 2015 Jul 9. PMID 26321369
- [Background] Krogh J, Gotze JP, Jorgensen MB, Kristensen LO, Kistorp C, Nordentoft M. Copeptin during rest and exercise in major depression. J Affect Disord. 2013 Oct;151(1):284-90. doi: 10.1016/j.jad.2013.06.007. Epub 2013 Jul 13. PMID 23856279
- [Background] Siegenthaler J, Walti C, Urwyler SA, Schuetz P, Christ-Crain M. Copeptin concentrations during psychological stress: the PsyCo study. Eur J Endocrinol. 2014 Dec;171(6):737-42. doi: 10.1530/EJE-14-0405. Epub 2014 Sep 23. PMID 25249697
- [Background] Kaczmarczyk M, Spitzer C, Wingenfeld K, Wiedemann K, Kuehl LK, Schultebraucks K, Deuter CE, Otte C. No association between major depression with and without childhood adversity and the stress hormone copeptin. Eur J Psychotraumatol. 2020 Nov 2;11(1):1837511. doi: 10.1080/20008198.2020.1837511. PMID 33244366
- [Background] Agorastos A, Sommer A, Heinig A, Wiedemann K, Demiralay C. Vasopressin Surrogate Marker Copeptin as a Potential Novel Endocrine Biomarker for Antidepressant Treatment Response in Major Depression: A Pilot Study. Front Psychiatry. 2020 May 20;11:453. doi: 10.3389/fpsyt.2020.00453. eCollection 2020. PMID 32508691
- [Derived] Milos Nymberg V, Pikkemaat M, Calling S, Nymberg P. HEAD-MIP-(HEAlth Dialogues for patients with Mental Illness in Primary care)-a feasibility study. Pilot Feasibility Stud. 2023 Sep 28;9(1):167. doi: 10.1186/s40814-023-01391-2. PMID 37770967
- [Derived] Pikkemaat M, Nymberg VM, Nymberg P. Structured assessment of modifiable lifestyle habits among patients with mental illnesses in primary care. Sci Rep. 2022 Jul 19;12(1):12292. doi: 10.1038/s41598-022-16439-1. PMID 35853972